CLINICAL TRIAL: NCT05702801
Title: Subsensory Stochastic Vibratory Stimulation to Assess and Improve Aging Related Proprioceptive Deficits Associated With Balance Recovery
Brief Title: Vibratory Stimulation to Improve Balance Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000207
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Fall; Fall Injury
Keywords: Balance recovery; stochastic stimulation intervention; Older adults

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exposure to stochastic vibratory stimulation (Experimental): All participants will be exposed to vibratory stimulations at different levels of 0Hz, 40Hz, and 80Hz.
  Interventions: Device: Stochastic Vibratory Stimulation (SVS)

INTERVENTIONS:
Device: Stochastic Vibratory Stimulation (SVS) — Investigators implement stochastic vibratory stimulation (SVS) to alter proprioceptive performance by increasing excitement of type Ia afferents in muscle spindles. Based on previous preliminary data, vibration frequencies around 40Hz may provide adequate noise for enhancing aging-related proprioceptive deficits. To make a subsensory noise investigators set it to 90% of the sensory threshold amplitude, which has been effectively used previously for influencing mechanoreceptor sensation in older adults. Stimulation will be imposed bilaterally on: 1) distal ankle (tibialis anterior, peroneus longus, soleus, gastrocnemius); and 2) proximal hip (quadriceps, gluteus medius, and paraspinals). Investigators use Gaussian noise to reduce the anticipative and preemptive adjustments of muscle spindles to the vibration. For SVS investigators use a magnetic actuator system and a Universal Controller (C-2HDLF Tactor/TDK), to provide programmable frequency ranges.

SUMMARY:
Falls are the primary cause of traumatic injury in older adults, and tripping is the leading cause of falls. A robust method for improving aging-related proprioceptive deficits is lacking, while strong evidence shows that proprioception deficits are highly associated with poor balance recovery from tripping. Previous research suggested that stochastic vibratory stimulation (SVS) can influence proprioception (i.e., muscle spindle function) among healthy controls; however, it is not clear how older adults with deficits in muscle spindle function would react to SVS. In previous work the investigators showed promising findings of standing balance and timed-up-and-go (TUG) improvements using SVS among high fall risk older adults with history of fall 15-18. They will implement SVS in the current project to improve aging-related proprioceptive deficits. The hypothesis is that SVS improves muscle spindle function and balance recovery from tripping in older adults with proprioceptive deficits.

DETAILED DESCRIPTION:
In this study investigators will assess the application of a novel methodology, stochastic vibratory stimulation (SVS), for enhancing proprioceptive performance in high fall risk older adults. It is hypothesized that SVS can alter muscle spindle activation. In high fall risk older adults, this additional activation effect on muscle spindle can improve deficits in proprioception. Two groups of low and high fall risk older adults, aged 65 and older, will be recruited. Both groups will go through several testing, including fall risk assessment, clinical questionnaires, proprioceptive measurement, and treadmill perturbation. Investigators will perform Stopping Elderly Accidents, Deaths & Injuries (STEADI) for fall screening, which includes: 1) fall history, unsteadiness, and fear of falling; 2) timed-up-and-go; 3) 30-second chair stand; and 4) four stage Romberg balance test. Questionnaires include: 1) fear of falling (Falls Efficacy Scale-International (FES-I)); 2) cognition (Montreal Cognitive Assessment - MoCA); 3) comorbidity (CMS Hierarchical Condition Category - CMS-HCC); 4) depression (Patient Health Questionnaire - PHQ-9); 5) pain in lower-extremity (Visual Analog Scale - VAS); and 6) vestibular-related symptoms (Dizziness Handicap Inventory - DHI). For proprioceptive measurement, investigators will assess joint position sense for ankle and hip with and without SVS. In both tests, participants perform the assessments in a safe platform. For the ankle joint, investigators will assess targeted angles of 5° and 10° plantarflexion and 5° dorsiflexion in random order. For the hip joint, participants will flex the trunk and be instructed to stop at 25, 50, and 75% of the range of motion in a random order. Further, both groups of participants will be exposed to low-speed treadmill perturbation (sudden backward treadmill movement to impose a trip-like disturbance) with and without SVS. During the perturbation, participants will be protected from falling using a secure harness. SVS will be applied to the ankle and hip muscles randomly in two separate sessions to influence proprioceptive performance from each of these sites. For the ankle joint SVS will be applied to tibialis anterior, peroneus longus, soleus, gastrocnemius, and for the hip joint it will be applied to quadriceps, gluteus medius, and paraspinals. In each session, after practicing and warming up twice at a slow treadmill speed (0.1m/s), each participant will go through six trials of perturbation within two bouts (0.35m/s), one with SVS and one without. To minimize the anticipation effect, one trial of forward belt movement will be randomly assigned (0.2m/s). All participants will be exposed to all testing conditions (ankle and hip SVS exposures). Investigators will measure balance recovery performance from the treadmill perturbation based on kinematics and muscle activity measures using wearable sensors. Kinematics outcomes will assess response time, recovery step execution, and lower-extremity and trunk motion during recovery. Assessment of muscle activity will provide insights regarding the onset of muscle activities during the balance recovery for tibialis anterior, peroneus longus, soleus, gastrocnemius, quadriceps, and paraspinals, using surface electromyography. Investigators will perform multivariable repeated measures analysis using mixed effects modeling to assess: 1) the effect of vibration area on each individual balance recovery outcome; and 2) the association between ankle (or hip) proprioceptive performance and ankle (or hip) SVS-imposed changes in balance recovery outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older
* the ability to understand study instructions.

Exclusion Criteria:

* disorders associated with severe motor and balance deficits, including stroke, Parkinson's disease, severe arthritis, lower-extremity amputation, spinal cord pathologies (e.g., spinal stenosis), and diabetes
* history of severe vestibular disorder such as bilateral vestibular hypofunction or poorly-compensated unilateral vestibular hypofunction, or Dizziness Handicap Inventory (DHI) > 40
* central nervous disease
* cognitive impairment (MoCA score<20)
* vision problems including cataract, presbyopia, and similar problems that can influence balance
* sedating medication or alcohol consumption within 24 hours.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Balance recovery outcomes | Baseline for with and without SVS conditions
  Investigators will extract outcomes treadmill perturbation. Failing to recover from the perturbation will be identified if the entire body weight is supported by the harness. Recoveries with integrated weight support greater than 5% of the weight × second will be classified as harness-assisted recoveries. All other recoveries will be considered successful and will be used for kinematics and muscle response analysis. Kinematics outcomes will assess response time, recovery step execution, and lower-extremity and trunk motion during recovery. Investigators will also assess muscle activities (from tibialis anterior, peroneus longus, soleus, gastrocnemius, quadriceps, and paraspinals).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States